CLINICAL TRIAL: NCT05567224
Title: Connecting Low-Income Adults to Primary Care After Inpatient Discharge
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, CARRIE FRY, Assistant Professor, Department of Health Policy, Vanderbilt University Medical Center
Other Study IDs: 221128
Record Dates: First submitted 2022-09-30; First posted 2022-10-05 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-02

CONDITIONS: Health Care Utilization; Health Care Seeking Behavior
Keywords: Health Care Costs; Hospitalizations; Emergency Department Use; Health Care Accessibility; Medicaid; Low-income populations
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pilot Group: This group of TennCare recipients will be referred to VUMC primary care services and will be allowed to utilize these services for at least two years. Those referred to VUMC primary care services will be those who belong to the two of state's three Medicaid Managed Care plans who have agreed to participate in this pilot.
  Interventions: Other: Access to primary care services
- Control Group: This group of TennCare recipients will not be referred to VUMC primary care services and will receive care as usual. Those not referred to VUMC primary care services will be those who belong to one of the state's three Medicaid Managed Care plans who has not agreed to participate in this pilot.

INTERVENTIONS:
Other: Access to primary care services — Those in the pilot group will be referred to primary care services and allowed to utilize them for at least two years. Primary care services include access to a primary care physician, medical management, and other tasks typically performed by a general practitioner. Those referred to primary care services will not have access to other VUMC outpatient services.
  Groups: Pilot Group

SUMMARY:
Healthcare systems and insurers have tried to reduce costs by improving the care and coordination provided to patients with high healthcare spending. Often termed, "hotspotting", these interventions seek to lower costs by reducing care provided in fragmented, high-cost settings, including the emergency department and inpatient settings, by addressing the social determinants of health and improving patients' access to lower-cost, ambulatory settings. Vanderbilt University Medical Center (VUMC), in collaboration with Tennessee's Medicaid agency (TennCare), is piloting a program to reduce costs and improve the quality of care provided to high-risk TennCare enrollees by referring them from inpatient settings to VUMC primary care services. This study seeks to evaluate this pilot by comparing outcomes between Medicaid patients referred to VUMC primary care services and similar Medicaid patients not referred to VUMC primary care services using data from surveys and administrative sources, including electronic health records and health insurance claims.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Currently enrolled in Tennessee's Medicaid Program (TennCare)
* Presenting in VUMC's inpatient setting
* Reporting no active relationship with a primary care doctor
* Lives in Davidson County, Tennessee, or a surrounding county

Exclusion Criteria:

* Patients discharged to a setting other than the community (e.g. to a Skilled Nursing Facility)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age 18 or older who are currently enrolled in Tennesee's Medicaid program (TennCare) and who are presenting in VUMC's inpatient setting, and who report no active relationship with a primary care doctor.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Number of Inpatient Admissions | 30, 60, 90, 180, and 360 days
  How many times the participant is hospitalized within the specified time period

SECONDARY OUTCOMES:
Number of Emergency Department Visits | 30, 60, 90, 180, and 360 days
  How many times the participant presents to the emergency department within the specified time period
Number of Primary Care Visits | 30, 60, 90, 180, and 360 days
  How many times the participant has seen a primary care physician within the specified time period
Average Health Care Spending | 30, 60, 90, 180, and 360 days
  Health care expenditures by the patient within the specified time frame
Average Self-reported Health Status | 30, 60, 90, 180, and 360 days
  A measure of the patient's self-reported physical and mental health, as measured by a shorter, modified version of the Short Form (SF)-36
Average of Disease Specific Outcomes | 30, 60, 90, 180, and 360 days
  Depending on the clinical information that is captured, disease specific clinical outcomes (e.g. prevalence of hypertension; HbA1C levels) will also be reported

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No